CLINICAL TRIAL: NCT03321435
Title: The Effect of Placenta Previa on Fetal Weight and Feto-maternal Blood Flow
Brief Title: The Placenta Previa and Fetal Weight
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: PPIUGR
Record Dates: First submitted 2017-10-21; First posted 2017-10-25 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- placenta previa group
  Interventions: Other: placenta previa patient
- Normal control group
  Interventions: Other: normal women

INTERVENTIONS:
Other: placenta previa patient — women had placenta previa either major or minor degree
  Groups: placenta previa group
Other: normal women — those women had not placenta previa
  Groups: Normal control group

SUMMARY:
Placenta previa is a placenta that implants at lower uterine segment, it occurs in about 0.3-0.5% of pregnancies at term. It is a significant risk for development of maternal morbidity, as well as maternal mortality secondary to maternal hemorrhage . Also, this abnormal placenta has a negative concern about fetal well being due to prematurity and perinatal mortality, in addition to its undesirable effect on fetal growth. Several factors may be behind of the effect of placenta previa on fetal growth. Firstly, the blood supply to the lower uterine segment is less than at the upper segment apparently resulting in less feto-placental blood perfusion . Secondly, recurrent bleeding attacks from placental previa may affect fetal oxygenation and fetal growth.

In spite of above evidences; many studies in literature denied the relation between placenta previa and fetal growth and concluded that the association between low birth weight and placenta previa is mainly due to preterm delivery and to a lesser extent with fetal growth restriction. However; the major drawback of all these studies is lacking of reporting the effect of placenta previa of feto-maternal blood flow representing in studying of Doppler blood flow in both uterine and umbilical artery in those patients. The uterine artery blood flow is usually affected by the presence of placenta previa and placenta accreta which reflected on feto-placental blood flow. So the uterine artery Doppler velocimetry is a useful tool for predicting placenta accreta .

So in the light of above evidences; we aimed, in the current study, not only to investigate the effect on placenta previa on fetal weight but also to walk around the effect of placenta previa on the uterine and umbilical arteries blood flow in trial to explore this conflicting issue. To our knowledge, no previous trial had studied this interesting subject before.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are sure of her pregnancy.
2. Women aged 20-35 years.
3. Women with BMI 18-22 kg/m2.
4. Estimated gestational age is ranging between 30- 32 weeks gestation.
5. Singleton pregnancy.
6. Placenta previa; either major or minor degrees as regard the cases.
7. Placenta previa with minimal vaginal bleeding or haven't any vaginal bleeding.
8. Women with normal Doppler indices in uterine and umbilical arteries at time of recruitment.
9. Women should be living in a nearby area to make follow-up and early transportation are reasonably possible.

Exclusion Criteria:

1. Women aged < 20 and >35 years.
2. Smoker ≥ 11 cigarettes/day.
3. Severe attack of bleeding requiring an immediate intervention.
4. Fetal heart rates instability or non reassuring.
5. Multiple gestations.
6. Previous Intrauterine growth restricted fetus.
7. Intrauterine fetal death or major fetal anomalies.
8. If associated with abruptio placentae.
9. Patients with known bleeding disorders or on anticoagulant therapy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: placenta previa patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Estimated fetal wight (gram) | 4 weeks

SECONDARY OUTCOMES:
The value of Doppler indices in uterine artery | 4 weeks